CLINICAL TRIAL: NCT03730389
Title: External Physical Vibration Lithecbole(EPVL) Versus Traditional Treatment for 4-10 mm Ureteral Stone: A Multi-center Prospective Randomized Controlled Trial
Brief Title: External Physical Vibration Lithecbole(EPVL) Versus Traditional Treatment for 4-10 mm Ureteral Stone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guohua Zeng (Other)
Responsible Party: Sponsor-Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPVL for 4-10mm ureteral stone
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Ureteral Calculi
Keywords: Ureteral Calculi; External Physical Vibration Lithecbole (EPVL); Efficacy; Safety
MeSH Terms: conditions — Ureteral Calculi

STUDY DESIGN:
Intervention Model Description: External Physical Vibration Lithecbole(EPVL) for ureteral stone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPVL Group (Experimental): In treatment group, patients were given one to three sessions of External Physical Vibration Lithecbole therapy in two weeks. These patients were also instructed to drink a minimum of 2500 ml water daily and take more exercise.
  Interventions: Device: External Physical Vibration Lithecbole (EPVL)
- Traditional Group (No Intervention): patients with 4-10mm ureteral stone, were treated by traditional treatment methods, including drinking a minimum of 2500 ml water daily and taking more exercise.

INTERVENTIONS:
Device: External Physical Vibration Lithecbole (EPVL) — Using the the way of external physical vibration to promote separation of stones from ureteral mucosa and promoting the excretion of ureteral stones
  Arms: EPVL Group

SUMMARY:
The investigator aims to perform a prospective and randomized controlled trial evaluating the safety and efficacy of External Physical Vibration Lithecbole(EPVL) in treating 4-10 mm ureteral stone.

DETAILED DESCRIPTION:
Patients with ureteral stones less than 10 mm, would receive observation for stone passage, not requiring immediate surgery. There are many studies evaluating the effect of Medical expulsive therapy in treating ureteral stones, including a-blockers, and calcium channel blockers. Most of shuties concluded that the benefit of a-blockers might be among those with larger (distal) stones. There is no good method for the removal of upper ureteral calculi, except drinking water and exercising.

Recently, a new extracorporeal physical vibrational lithecbole (EPVL) device named Friend-I EPVL (Zhengzhou Fu Jian Da Medical Instrument Co., Zhengzhou, China) has proven to be an effective treatment for upper urinary tract residual calculi. The device was approved by the Chinese food and drug administration in 2012. A Simple harmonic motion technology in multi-direction was applied. The Lateral acceleration was provided by the physical vibration device in the base through the harmonic vibration wave in the horizontal direction, which induces the urinary stone separate with the kidney or ureter, and expands a moving space for the stone. Meanwhile, an axial effect was produced to push the stone by the physical vibration device in the handle through the harmonic vibration wave in the multi- direction. So, we think that EPVL may be effective in treating ureteral stones.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 to 70 years
2. 4-10 mm single ureteral calculi
3. Normal serum creatinine
4. ASA grading: 1-2 levels.

Exclusion Criteria:

1. Pregnant or isolated kidney patients
2. Moderate or severe hydronephrosis
3. History of ureteral stricture
4. Multiple ureteral stones;
5. Acute urinary tract infection
6. Those who are taking α-receptor, calcium channel blocker or chinese medicine stone shovel
7. Dysfunction of blood coagulation
8. Obese patients (body mass index > 28 kg / m2);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Stone Expulsion | 14 days
  The stone discharge rate of the two group

SECONDARY OUTCOMES:
Time to Stone Passage | 14 days
  Time to stone elimination in days in patients with spontaneous elimination
The rate of renal colic | 14 days
  the mean rate of renal colic between the two groups
Required Analgesics | 14 days
  the need for slow-released diclofenac tablet

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D & MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No